CLINICAL TRIAL: NCT02176135
Title: A Dose Escalation Phase I Study to Evaluate the Safety and Tolerability of Oral Auranofin Therapy in HIV-infected Subjects Receiving Suppressive Antiretroviral Therapy
Brief Title: Oral Auranofin for Reduction of Latent Viral Reservoir in Patients With HIV Infection
Acronym: Goldrake
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vaccine and Gene Therapy Institute, Florida (Other)
Collaborators: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUR-001
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: HIV
Keywords: HIV; HAART suppressed; Auranofin; HIV latent reservoir
MeSH Terms: interventions — Auranofin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose escalation (Experimental): Auranofin 3 to 6 mg/day oral administration for 12 weeks
  Interventions: Drug: Auranofin

INTERVENTIONS:
Drug: Auranofin — 3 mg tablets
  Other Names: Ridaura

SUMMARY:
The main purpose of the study is to evaluate the safety of oral auranofin, a gold compound, in patients with HIV infection whose viral load has been suppressed by antiretroviral therapy for no less than 3 years and have a CD4+ cell count over 500 cells/uL

DETAILED DESCRIPTION:
The investigators proposed a novel approach in order to reduce the HIV viral reservoir. This approach exploits the effects of auranofin, a gold based compound which has been used in the treatment of rheumatoid arthritis. Auranofin induces partially selective apoptosis and differentiation towards short-lived phenotypes of the T lymphocyte memory subsets that encompass the main viral reservoir in patients. The hypothesis is that the targeted memory cells would either die or decrease their persistence in the body, with the associated latent viral reservoir being reduced.

The study will be conducted in two phases: A sequential dose-escalation phase to evaluate two doses of auranofin, followed by an expansion at the maximum tolerated dose (MTD). A total of 20 patients are to be treated at the MTD. Auranofin treatment is administered for 12 weeks.

Safety and tolerability will be evaluated by repeated laboratory panel and physcial examination during the 12 weeks of auranofin therapy and 8 for weeks thereafter. The latent reservoir will be measured by assessment of the inegrated viral DNA in CD4+ cells in the circulating blood and in gut biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or female, between 18 and 55 years of age.
* Stable dose of ART (defined as at least 2 nucleoside/nucleotide reverse transcriptase inhibitors plus a non-nucleoside reverse transcriptase inhibitor, integrase inhibitor, or a protease inhibitor) for at least 2 years from study consent and with no modifications expected during the study.
* HIV plasma viral load <50 copies/ml for at least 3 years with several measurements per year and most recent viral load within 3 months of screening.8
* No previous failure of ART, understood as a rebound in viral load that can be detected after having reached undetectable levels. Low-grade increases (<200 copies of HIV RNA/mL) and transitory increases (blips) resolved without modifying ART are acceptable.
* Did not experience AIDS defining event
* Two CD4+ T cell counts greater than 500 cell/µl in the six months prior to screening
* Able (in the Investigators' opinion) and willing to comply with all study requirements.

Exclusion Criteria:

* Contraindication to auranofin therapy, including congestive heart failure, renal dysfunction, history of blood dyscrasias; History of gold induced disorders (e.g. necrotising enterocolitis, pulmonary fibrosis, exfoliative dermatitis, bone marrow aplasia or other sever hematologic disorders), porphyria; History of severe allergic or anaphylactic reactions or hypersensitivity to auranofin or other gold compounds.
* Treatment with nucleoside/nucleotide analogs with higher risk of mitochondrial toxicity: zidovudine (ZDV), Stavudine (d4T), didanosine (ddI), di-deoxy-cytidine (ddC) or abacavir (ABC).
* Presence of clinically significant skin/mucosal disease such as hives or dermatitis, pruritus or rash, eczema, stomatitis or conjunctivitis
* Significant acute medical illness in the past 4 weeks
* Inflammatory bowel disease, Crohn's disease or ulcerative colitis
* Current or recent (i.e. within 2 weeks) gastrointestinal disease or GI disturbances, including vomiting, abdominal pain, diarrhea, which may impact the absorption of the investigational drug
* History of gastrointestinal surgery that could impact upon the absorption of Auranofin
* Scheduled elective surgery or other procedures requiring general anesthesia during the study
* Participant has the following laboratory values within 2 weeks before starting the investigational drug (laboratory tests may be repeated, as clinically indicated, to obtain acceptable values before failure at screening is concluded)
* Known hepatitis B or C infection as indicated by the presence of Hepatitis B surface antigen (HBsAg) or hepatitis C virus RNA (HCV-RNA) in blood
* Receipt of immunomodulating therapy, EPO or G-CSF, immunization or systemic chemotherapeutic agents within 12 weeks prior to study entry
* Anticipated requirement for treatment with drugs that may interfere with auranofin as outlined in Appendix 7.
* Receipt of RBC or platelet transfusion or receipt of cell product within 24 weeks prior to study entry
* Insulin dependent diabetes
* Systemic Lupus Erythematosus (SLE)
* Current or history of seizure disorder
* Previous diagnosis of lymphoma or other HIV related cancers.
* Any other significant disease or disorder (including psychiatric disorders) which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Women who are pregnant or breastfeeding, or with a positive pregnancy test during screening or Women of Child Bearing Potential (WOCBP) who are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for the entire study period and for at least 4 weeks before and 24 weeks after study treatment
* Males or females who are unwilling or unable to use barrier contraception during sexual intercourse for the entire study period, including at least 4 weeks before, 4 weeks after study treatment, and when plasma HIV-RNA is detectable using standard assays
* Subjects who have participated in another research study involving an investigational product in the past 12 weeks.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 12 weeks treatment and 8 weeks post-therapy
  Adverse event frequency and severity per NIAID ACTG grading tables

SECONDARY OUTCOMES:
Change from baseline in measures of the HIV latent reservoir during auranofin therapy | 12 weeks therapy and 8 weeks post-therapy
  The size of the latent reservoir will be measured by the frequency of CD4+ T cells harboring total and integrated HIV DNA and by the frequency of CD4+ T-cells cells harboring inducible HIV multiply-spliced RNA upon maximal stimulation (expressed as infected cells per million CD4+ T cells).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick D Yeramian, MD, Study Director — Vaccine and Gene Therapy Institute, Florida
Locations (1):
- University of Miami - AIDS Clinical Research Unit, Miami, Florida, United States